CLINICAL TRIAL: NCT06500377
Title: A Pilot Study Exploring Four Types of Meditation Practices for Relaxation Among Cancer Survivors
Brief Title: Comparing the Impact of Four Types of Meditation Practices for Relaxation in Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22607; NCI-2024-04827 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22607 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Arm I (breathing only meditation) (Experimental): Patients learn breathing only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Meditation Therapy; Other: Questionnaire Administration
- Arm I (focused attention only meditation) (Experimental): Patients learn focused attention only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Meditation Therapy; Other: Questionnaire Administration
- Arm III (mindfulness only meditation) (Experimental): Patients learn mindfulness only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Meditation Therapy; Other: Questionnaire Administration
- Arm IV (combined meditation) (Experimental): Patients learn breathing, focused attention, and mindfulness combined meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Meditation Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo saliva sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Meditation Therapy — Learn breathing only meditation
  Other Names: Meditation
  Arms: Arm I (breathing only meditation)
Procedure: Meditation Therapy — Learn focused attention only meditation
  Other Names: Meditation
  Arms: Arm I (focused attention only meditation)
Procedure: Meditation Therapy — Learn mindfulness only meditation
  Other Names: Meditation
  Arms: Arm III (mindfulness only meditation)
Procedure: Meditation Therapy — Learn breathing, focused attention, and mindfulness combined meditation
  Other Names: Meditation
  Arms: Arm IV (combined meditation)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares the impact of four types of meditation practices, breathing only, focused attention only, mindfulness only, and breathing, focused attention and mindfulness combined, for relaxation in cancer survivors. Studies show that many patients with cancer experience stress and anxiety. Meditation therapy uses a variety of techniques, such as breathing, sound, or movement, that may help to decrease distress and anxiety and enhance the health and quality of life of patients with cancer. The trial is being done to find out how meditation can help cancer survivors feel relaxed and attain a peaceful state of mind.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the feasibility to attend and complete the meditation program as scheduled (combined arms) within six weeks.

EXPLORATORY OBJECTIVES:

I. Assess the ability of breathing, mindfulness, focused attention, and a combination of all three meditation techniques to enhance relaxation in cancer survivors.

II. Determine which meditation technique improves the outcome measures the most.

III. Explore which meditation method is preferred by the subjects.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients learn breathing only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.

ARM II: Patients learn focused attention only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.

ARM III: Patients learn mindfulness only meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.

ARM IV: Patients learn breathing, focused attention, and mindfulness combined meditation with an instructor over 60 minutes for 3 sessions within 6 weeks. Patients also practice meditation at home and undergo saliva sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant
* Age: ≥ 18 years
* Ability to understand and fluently speak English or Spanish
* No previous training in mind-body relaxation techniques including meditation, yoga, tai chi, qigong, guided imagery, mindfulness-based stress reduction, hypnosis, or cognitive behavior therapy, that exceeds 3 hours. Additionally, no regular practice of mind-body relaxation techniques, or formal experience with mind-body relaxation techniques within the past 12 months
* Visual Analog Scale (VAS) anxiety score of > 3 from a range from 0 to 10. A "0" means the lowest anxiety score and a "10" means the highest anxiety score
* Long-term cancer survivors who received surgery to treat their cancer ( > 6 months since last treatment) with no history of chemotherapy, radiation therapy, or other systemic therapy (e.g., hormonal therapy) and/or have completely recovered from surgery OR patients identified as having pre-cancerous lesions that have been surgically treated (e.g., colon polyp that has been removed)
* Willingness to:

  * Provide salivary alpha-amylase sample
  * Complete stress tests and study questionnaires
  * Be monitored with a Bispectral Index (BIS) device

Exclusion Criteria:

* Inability to complete study required time and procedures as outlined in the study procedures section of the protocol
* Must not have had previous serious illnesses that affect neurological functioning such as strokes, heart attacks, Parkinson disease, etc
* Ongoing active psychiatric condition, depressive/bi-polar related disorders, anxiety, psychosis disorders, or substance use that may interfere with the study including panic disorder, major depression, schizophrenia, and bipolar disease
* Active cancer
* Cancer survivors who have received chemotherapy, radiation therapy, or any other systemic treatment (e.g., hormonal therapy)
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Retention rate | Up to 6 weeks
  Feasibility will be achieved if 70% of all enrolled participants attend at least 5 full visits within 6 weeks. Descriptive statistics will be generated.
Adherence rate | Up to 6 weeks
  Feasibility will be achieved if 70% of all enrolled participants complete all assessments of the program within 6 weeks. Descriptive statistics will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California